CLINICAL TRIAL: NCT05280158
Title: Phase I/II, Open-Label Dose-Finding Trial of High-Dose mRNA-1273 Booster for Lung Transplant Recipients
Brief Title: High-Dose Moderna mRNA-1273 Booster Study for Lung Transplant Recipients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Moderna Bivalent COVID-19 Vaccine became available to the public in Sept 2022.
Sponsor: University of California, Los Angeles (Other)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Y. Shino, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-000192
Record Dates: First submitted 2022-03-05; First posted 2022-03-15 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Lung Transplant Recipient; SARS-CoV-2; Immunosuppression
Keywords: SARS-CoV-2; lung transplant recipient; immunosuppression
MeSH Terms: interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Groups will be enrolled as follows:
  1. Mid-dose - Sentinel group, n=2
  2. Standard-dose - Initial group, n=2
  3. Cohort 1: 2:1 Randomization into
     * Mid-dose group, n=18
     * Standard-dose group, n=9
  4. High-dose - Sentinel group, n=2
  5. Cohort 2: 2:1 Randomization into
     * High-dose group, n=18
     * Standard-dose group, n=9
  We will perform stratified randomization for the two cohorts based on: 1) the number of prior doses, and 2) prior receipt of any BNT162b2 vaccines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard-dose (Active Comparator): mRNA-1273 (Moderna COVID-19 vaccine) 50 ug
  Interventions: Drug: mRNA-1273 (Moderna COVID-19 vaccine)
- Mid-Dose (Experimental): mRNA-1273 (Moderna COVID-19 vaccine) 100 ug
  Interventions: Drug: mRNA-1273 (Moderna COVID-19 vaccine)
- High-Dose (Experimental): mRNA-1273 (Moderna COVID-19 vaccine) 200 ug
  Interventions: Drug: mRNA-1273 (Moderna COVID-19 vaccine)

INTERVENTIONS:
Drug: mRNA-1273 (Moderna COVID-19 vaccine) — Study Drug will be administered via intramuscular injection (IM). Only one dose of study drug will be administered for the study.

SUMMARY:
Lung transplant recipients have poor outcomes after COVID-19 infection with mortality. Due to the immunosuppression, they have had poor responses to SARS-CoV-2 vaccine and remain at high risk of poor outcomes. This is a Phase I/II clinical trial to evaluate the safety and immune response from a higher dose mRNA-1273 vaccine among lung transplant recipients who have already received three or four doses of the COVID-19 vaccine.

DETAILED DESCRIPTION:
This is a Phase I/II open-label dose-finding trial among lung transplant recipients who received three or four mRNA vaccine doses (mRNA-1273 or BNT162b2) after lung transplantation to: standard-dose (50 ug), mid-dose (100 ug) or high-dose (200 ug) mRNA-1273 booster vaccine. Sixty participants will be enrolled into three dose groups: 1) Standard-dose - 20 participants, 2) Mid-dose - 20 participants, 3) High-dose - 20 participants. The first 2 participants in both the mid-dose and high dose groups will be considered the 'sentinel' group. Participants in the sentinel group will receive the vaccine and undergo a 7-day observation period for safety and reactogenicity before additional participants are enrolled into that dose group.

Overall study enrollment will begin with the mid-dose sentinel group (n=2). During the observation period for the mid-dose sentinel group, we will enroll two participants into the standard-dose group. Once the mid-dose sentinel group completes their 7-day observation period without triggering halting rules and is approved to proceed by the DSMB, we will enroll the next 27 participants (Cohort 1) with a 2:1 randomization into the mid-dose (n=18) and standard-dose (n=9) groups.

Once all 20 participants have received their mid-dose vaccine without triggering halting rules and is approved to proceed by the DSMB, we will enroll the high-dose sentinel group (n=2). Once the high-dose sentinel group completes their 7-day observation period without triggering halting rules and is approved to proceed by the DSMB, we will enroll the next 27 participants (Cohort 2) with a 2:1 randomization into the high-dose (n=18) and standard-dose (n=9) groups. All 20 participants in the mid-dose group will be enrolled prior to the enrollment of the high-dose group.

We will perform stratified randomization for the two cohorts based on: 1) the number of prior doses, and 2) prior receipt of any BNT162b2 vaccines. Randomization with be done by the UCLA Clinical and Translational Science Institute (CTSI) statistics team based on scheduled participants prior to the study visit. The 6 participants in the sentinel (n=4) and initial (n=2) groups (Table 1) will be assigned into the 3 groups based on their scheduled visit day.

ELIGIBILITY:
1. All adult lung transplant recipients (age ≥ 18 at the time of consent) who received all of their COVID-19 vaccines after lung transplantation.
2. Received three or four doses of either the Moderna mRNA-1273 or Pfizer BNT162b2 vaccine with the last dose received at least 4 months prior to study enrollment.
3. Currently receiving standard regimen of three drug immunosuppression with prednisone, tacrolimus and mycophenolate mofetil (cellcept, minimum 250 mg bid) or mycophenolate sodium (myfortic, minimum 180 mg bid).
4. Agrees not to receive other investigational agents for prophylaxis against COVID-19 including Evusheld monoclonal antibodies for at least 30 days after the study vaccine.
5. Understands and agrees to comply with the study procedures and provides written informed consent.
6. Is in stable health without any new or worsening medical conditions in the opinion of the Investigator.
7. Female participants of childbearing potential (<1 year since start of menopause) may be enrolled in the study if the participant fulfills all the following criteria:

   1. Has a negative pregnancy test at Visit 1 Day 1.
   2. Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection (Day 1).
   3. Has agreed to continue adequate contraception or practice abstinence through 3 months following the booster injection (Day 90).
   4. Is not currently breastfeeding.
   5. Adequate female contraception is defined as consistent and correct use of a Food and Drug Administration (FDA) approved contraceptive method in accordance with the product label. For example:

   i. Barrier method (such as condoms, diaphragm, or cervical cap) used in conjunction with spermicide ii. Intrauterine device iii. Prescription hormonal contraceptive taken or administered via oral (pill), transdermal (patch), subdermal, or IM route iv. Sterilization of a female participant's monogamous male partner prior to entry into the study v. Note: periodic abstinence (e.g., calendar, ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Previous documented COVID-19 infection.
2. Use of investigational agents for prophylaxis against COVID-19 within 90 days of the start of the study, including Evusheld monoclonal antibodies.
3. Ongoing therapy for acute cellular or antibody mediated rejection.
4. Intravenous immunoglobulins (IVIG) administration within the prior 3 months or ongoing IVIG therapy.
5. Anaphylaxis or allergic reaction to any prior vaccines.
6. History of anaphylaxis or other significant adverse reaction requiring medical intervention after receipt of a vaccine.
7. Is acutely ill or febrile 24 hours prior to or at the Day 1 visit. Fever is defined as a body temperature ≥ 38.0°C/100.4°F. Participants meeting this criterion may be rescheduled within the relevant window periods. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
8. Pregnant or breastfeeding.
9. Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
10. Known history of hypertension (HTN) with systolic blood pressure (BP) > 180 mm Hg at the Day 1 visit.
11. Known history of hypotension with systolic blood pressure < 85 mm Hg at the Day 1 visit.
12. Bleeding disorder considered a contraindication to IM injection or phlebotomy.
13. Active malignancy diagnosed within previous 4 years (excluding non-melanoma skin cancer).
14. Received a major surgery including lung transplantation in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusaku Michael Shino, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Clinical Translational Research Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corbett KS, Flynn B, Foulds KE, Francica JR, Boyoglu-Barnum S, Werner AP, Flach B, O'Connell S, Bock KW, Minai M, Nagata BM, Andersen H, Martinez DR, Noe AT, Douek N, Donaldson MM, Nji NN, Alvarado GS, Edwards DK, Flebbe DR, Lamb E, Doria-Rose NA, Lin BC, Louder MK, O'Dell S, Schmidt SD, Phung E, Chang LA, Yap C, Todd JM, Pessaint L, Van Ry A, Browne S, Greenhouse J, Putman-Taylor T, Strasbaugh A, Campbell TA, Cook A, Dodson A, Steingrebe K, Shi W, Zhang Y, Abiona OM, Wang L, Pegu A, Yang ES, Leung K, Zhou T, Teng IT, Widge A, Gordon I, Novik L, Gillespie RA, Loomis RJ, Moliva JI, Stewart-Jones G, Himansu S, Kong WP, Nason MC, Morabito KM, Ruckwardt TJ, Ledgerwood JE, Gaudinski MR, Kwong PD, Mascola JR, Carfi A, Lewis MG, Baric RS, McDermott A, Moore IN, Sullivan NJ, Roederer M, Seder RA, Graham BS. Evaluation of the mRNA-1273 Vaccine against SARS-CoV-2 in Nonhuman Primates. N Engl J Med. 2020 Oct 15;383(16):1544-1555. doi: 10.1056/NEJMoa2024671. Epub 2020 Jul 28. PMID 32722908
- [Background] Corbett KS, Nason MC, Flach B, Gagne M, O'Connell S, Johnston TS, Shah SN, Edara VV, Floyd K, Lai L, McDanal C, Francica JR, Flynn B, Wu K, Choi A, Koch M, Abiona OM, Werner AP, Moliva JI, Andrew SF, Donaldson MM, Fintzi J, Flebbe DR, Lamb E, Noe AT, Nurmukhambetova ST, Provost SJ, Cook A, Dodson A, Faudree A, Greenhouse J, Kar S, Pessaint L, Porto M, Steingrebe K, Valentin D, Zouantcha S, Bock KW, Minai M, Nagata BM, van de Wetering R, Boyoglu-Barnum S, Leung K, Shi W, Yang ES, Zhang Y, Todd JM, Wang L, Alvarado GS, Andersen H, Foulds KE, Edwards DK, Mascola JR, Moore IN, Lewis MG, Carfi A, Montefiori D, Suthar MS, McDermott A, Roederer M, Sullivan NJ, Douek DC, Graham BS, Seder RA. Immune correlates of protection by mRNA-1273 vaccine against SARS-CoV-2 in nonhuman primates. Science. 2021 Sep 17;373(6561):eabj0299. doi: 10.1126/science.abj0299. Epub 2021 Sep 17. PMID 34529476
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] El Sahly HM, Baden LR, Essink B, Doblecki-Lewis S, Martin JM, Anderson EJ, Campbell TB, Clark J, Jackson LA, Fichtenbaum CJ, Zervos M, Rankin B, Eder F, Feldman G, Kennelly C, Han-Conrad L, Levin M, Neuzil KM, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Polakowski L, Mascola JR, Ledgerwood JE, Graham BS, August A, Clouting H, Deng W, Han S, Leav B, Manzo D, Pajon R, Schodel F, Tomassini JE, Zhou H, Miller J; COVE Study Group. Efficacy of the mRNA-1273 SARS-CoV-2 Vaccine at Completion of Blinded Phase. N Engl J Med. 2021 Nov 4;385(19):1774-1785. doi: 10.1056/NEJMoa2113017. Epub 2021 Sep 22. PMID 34551225
- [Background] Oliver SE, Wallace M, See I, Mbaeyi S, Godfrey M, Hadler SC, Jatlaoui TC, Twentyman E, Hughes MM, Rao AK, Fiore A, Su JR, Broder KR, Shimabukuro T, Lale A, Shay DK, Markowitz LE, Wharton M, Bell BP, Brooks O, McNally V, Lee GM, Talbot HK, Daley MF. Use of the Janssen (Johnson & Johnson) COVID-19 Vaccine: Updated Interim Recommendations from the Advisory Committee on Immunization Practices - United States, December 2021. MMWR Morb Mortal Wkly Rep. 2022 Jan 21;71(3):90-95. doi: 10.15585/mmwr.mm7103a4. PMID 35051137
- [Background] Barda N, Dagan N, Ben-Shlomo Y, Kepten E, Waxman J, Ohana R, Hernan MA, Lipsitch M, Kohane I, Netzer D, Reis BY, Balicer RD. Safety of the BNT162b2 mRNA Covid-19 Vaccine in a Nationwide Setting. N Engl J Med. 2021 Sep 16;385(12):1078-1090. doi: 10.1056/NEJMoa2110475. Epub 2021 Aug 25. PMID 34432976
- [Background] Simone A, Herald J, Chen A, Gulati N, Shen AY, Lewin B, Lee MS. Acute Myocarditis Following COVID-19 mRNA Vaccination in Adults Aged 18 Years or Older. JAMA Intern Med. 2021 Dec 1;181(12):1668-1670. doi: 10.1001/jamainternmed.2021.5511. PMID 34605853
- [Background] Oster ME, Shay DK, Su JR, Gee J, Creech CB, Broder KR, Edwards K, Soslow JH, Dendy JM, Schlaudecker E, Lang SM, Barnett ED, Ruberg FL, Smith MJ, Campbell MJ, Lopes RD, Sperling LS, Baumblatt JA, Thompson DL, Marquez PL, Strid P, Woo J, Pugsley R, Reagan-Steiner S, DeStefano F, Shimabukuro TT. Myocarditis Cases Reported After mRNA-Based COVID-19 Vaccination in the US From December 2020 to August 2021. JAMA. 2022 Jan 25;327(4):331-340. doi: 10.1001/jama.2021.24110. PMID 35076665
- [Background] Larson KF, Ammirati E, Adler ED, Cooper LT Jr, Hong KN, Saponara G, Couri D, Cereda A, Procopio A, Cavalotti C, Oliva F, Sanna T, Ciconte VA, Onyango G, Holmes DR, Borgeson DD. Myocarditis After BNT162b2 and mRNA-1273 Vaccination. Circulation. 2021 Aug 10;144(6):506-508. doi: 10.1161/CIRCULATIONAHA.121.055913. Epub 2021 Jun 16. PMID 34133884
- [Background] Rosenblum HG, Hadler SC, Moulia D, Shimabukuro TT, Su JR, Tepper NK, Ess KC, Woo EJ, Mba-Jonas A, Alimchandani M, Nair N, Klein NP, Hanson KE, Markowitz LE, Wharton M, McNally VV, Romero JR, Talbot HK, Lee GM, Daley MF, Mbaeyi SA, Oliver SE. Use of COVID-19 Vaccines After Reports of Adverse Events Among Adult Recipients of Janssen (Johnson & Johnson) and mRNA COVID-19 Vaccines (Pfizer-BioNTech and Moderna): Update from the Advisory Committee on Immunization Practices - United States, July 2021. MMWR Morb Mortal Wkly Rep. 2021 Aug 13;70(32):1094-1099. doi: 10.15585/mmwr.mm7032e4. PMID 34383735
- [Background] Marion O, Del Bello A, Abravanel F, Couat C, Faguer S, Esposito L, Hebral AL, Izopet J, Kamar N. Safety and Immunogenicity of Anti-SARS-CoV-2 Messenger RNA Vaccines in Recipients of Solid Organ Transplants. Ann Intern Med. 2021 Sep;174(9):1336-1338. doi: 10.7326/M21-1341. Epub 2021 May 25. No abstract available. PMID 34029487
- [Background] Hall VG, Ferreira VH, Ku T, Ierullo M, Majchrzak-Kita B, Chaparro C, Selzner N, Schiff J, McDonald M, Tomlinson G, Kulasingam V, Kumar D, Humar A. Randomized Trial of a Third Dose of mRNA-1273 Vaccine in Transplant Recipients. N Engl J Med. 2021 Sep 23;385(13):1244-1246. doi: 10.1056/NEJMc2111462. Epub 2021 Aug 11. No abstract available. PMID 34379917
- [Background] Boyarsky BJ, Werbel WA, Avery RK, Tobian AAR, Massie AB, Segev DL, Garonzik-Wang JM. Antibody Response to 2-Dose SARS-CoV-2 mRNA Vaccine Series in Solid Organ Transplant Recipients. JAMA. 2021 Jun 1;325(21):2204-2206. doi: 10.1001/jama.2021.7489. PMID 33950155
- [Background] Schramm R, Costard-Jackle A, Rivinius R, Fischer B, Muller B, Boeken U, Haneya A, Provaznik Z, Knabbe C, Gummert J. Poor humoral and T-cell response to two-dose SARS-CoV-2 messenger RNA vaccine BNT162b2 in cardiothoracic transplant recipients. Clin Res Cardiol. 2021 Aug;110(8):1142-1149. doi: 10.1007/s00392-021-01880-5. Epub 2021 Jul 9. PMID 34241676
- [Background] Shostak Y, Shafran N, Heching M, Rosengarten D, Shtraichman O, Shitenberg D, Amor SM, Yahav D, Ben Zvi H, Pertzov B, Kramer MR. Early humoral response among lung transplant recipients vaccinated with BNT162b2 vaccine. Lancet Respir Med. 2021 Jun;9(6):e52-e53. doi: 10.1016/S2213-2600(21)00184-3. Epub 2021 May 5. No abstract available. PMID 33964244
- [Background] Havlin J, Svorcova M, Dvorackova E, Lastovicka J, Lischke R, Kalina T, Hubacek P. Immunogenicity of BNT162b2 mRNA COVID-19 vaccine and SARS-CoV-2 infection in lung transplant recipients. J Heart Lung Transplant. 2021 Aug;40(8):754-758. doi: 10.1016/j.healun.2021.05.004. Epub 2021 May 21. PMID 34120839
- [Background] Messika J, Eloy P, Roux A, Hirschi S, Nieves A, Le Pavec J, Senechal A, Saint Raymond C, Carlier N, Demant X, Le Borgne A, Tissot A, Debray MP, Beaumont L, Renaud-Picard B, Reynaud-Gaubert M, Mornex JF, Falque L, Boussaud V, Jougon J, Mussot S, Mal H; French Group of Lung Transplantation. COVID-19 in Lung Transplant Recipients. Transplantation. 2021 Jan 1;105(1):177-186. doi: 10.1097/TP.0000000000003508. PMID 33141808
- [Background] Saez-Gimenez B, Berastegui C, Barrecheguren M, Revilla-Lopez E, Los Arcos I, Alonso R, Aguilar M, Mora VM, Otero I, Reig JP, Quezada CA, Perez V, Valle M, Laporta R, Deu M, Sacanell J, Bravo C, Gavalda J, Lopez-Meseguer M, Monforte V. COVID-19 in lung transplant recipients: A multicenter study. Am J Transplant. 2021 May;21(5):1816-1824. doi: 10.1111/ajt.16364. Epub 2020 Nov 7. PMID 33089648
- [Background] Aversa M, Benvenuto L, Anderson M, Shah L, Robbins H, Pereira M, Scheffert J, Carroll M, Hum J, Nolan M, Reilly G, Lemaitre P, Stanifer BP, D'Ovidio F, Sonett J, Arcasoy S; From the Columbia University Lung Transplant Program. COVID-19 in lung transplant recipients: A single center case series from New York City. Am J Transplant. 2020 Nov;20(11):3072-3080. doi: 10.1111/ajt.16241. Epub 2020 Sep 5. PMID 32881315
- [Background] Kamp JC, Hinrichs JB, Fuge J, Ewen R, Gottlieb J. COVID-19 in lung transplant recipients-Risk prediction and outcomes. PLoS One. 2021 Oct 6;16(10):e0257807. doi: 10.1371/journal.pone.0257807. eCollection 2021. PMID 34613977
- [Background] Hall VG, Ferreira VH, Ierullo M, Ku T, Marinelli T, Majchrzak-Kita B, Yousuf A, Kulasingam V, Humar A, Kumar D. Humoral and cellular immune response and safety of two-dose SARS-CoV-2 mRNA-1273 vaccine in solid organ transplant recipients. Am J Transplant. 2021 Dec;21(12):3980-3989. doi: 10.1111/ajt.16766. Epub 2021 Aug 4. PMID 34347934
- [Background] Kamar N, Abravanel F, Marion O, Couat C, Izopet J, Del Bello A. Three Doses of an mRNA Covid-19 Vaccine in Solid-Organ Transplant Recipients. N Engl J Med. 2021 Aug 12;385(7):661-662. doi: 10.1056/NEJMc2108861. Epub 2021 Jun 23. No abstract available. PMID 34161700
- [Background] Werbel WA, Boyarsky BJ, Ou MT, Massie AB, Tobian AAR, Garonzik-Wang JM, Segev DL. Safety and Immunogenicity of a Third Dose of SARS-CoV-2 Vaccine in Solid Organ Transplant Recipients: A Case Series. Ann Intern Med. 2021 Sep;174(9):1330-1332. doi: 10.7326/L21-0282. Epub 2021 Jun 15. No abstract available. PMID 34125572
- [Background] Damluji AA, Christenson RH, deFilippi C. Clinical Application of Serologic Testing for Coronavirus Disease 2019 in Contemporary Cardiovascular Practice. J Am Heart Assoc. 2021 Feb;10(5):e019506. doi: 10.1161/JAHA.120.019506. Epub 2021 Feb 23. PMID 33619984
- [Background] Abu S, Roguin A, Hellou E, Ishai A, Shoshan U, Mahamid L. Since January 2020 Elsevier has created a COVID-19 resource centre with free information in English and Mandarin on the novel coronavirus COVID- 19 . The COVID-19 resource centre is hosted on Elsevier Connect , the company ' s public news and information . 2020;
- [Background] Patone M, Mei XW, Handunnetthi L, Dixon S, Zaccardi F, Shankar-Hari M, Watkinson P, Khunti K, Harnden A, Coupland CAC, Channon KM, Mills NL, Sheikh A, Hippisley-Cox J. Risks of myocarditis, pericarditis, and cardiac arrhythmias associated with COVID-19 vaccination or SARS-CoV-2 infection. Nat Med. 2022 Feb;28(2):410-422. doi: 10.1038/s41591-021-01630-0. Epub 2021 Dec 14. PMID 34907393
- [Background] Gargano JW, Wallace M, Hadler SC, Langley G, Su JR, Oster ME, Broder KR, Gee J, Weintraub E, Shimabukuro T, Scobie HM, Moulia D, Markowitz LE, Wharton M, McNally VV, Romero JR, Talbot HK, Lee GM, Daley MF, Oliver SE. Use of mRNA COVID-19 Vaccine After Reports of Myocarditis Among Vaccine Recipients: Update from the Advisory Committee on Immunization Practices - United States, June 2021. MMWR Morb Mortal Wkly Rep. 2021 Jul 9;70(27):977-982. doi: 10.15585/mmwr.mm7027e2. PMID 34237049
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455
- [Background] Aretz HT. Myocarditis: the Dallas criteria. Hum Pathol. 1987 Jun;18(6):619-24. doi: 10.1016/s0046-8177(87)80363-5. No abstract available. PMID 3297992
- [Background] Adler Y, Charron P, Imazio M, Badano L, Baron-Esquivias G, Bogaert J, Brucato A, Gueret P, Klingel K, Lionis C, Maisch B, Mayosi B, Pavie A, Ristic AD, Sabate Tenas M, Seferovic P, Swedberg K, Tomkowski W; ESC Scientific Document Group. 2015 ESC Guidelines for the diagnosis and management of pericardial diseases: The Task Force for the Diagnosis and Management of Pericardial Diseases of the European Society of Cardiology (ESC)Endorsed by: The European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2015 Nov 7;36(42):2921-2964. doi: 10.1093/eurheartj/ehv318. Epub 2015 Aug 29. No abstract available. PMID 26320112

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: High Dose arm was not recorded because no participants enrolled in this group.
Groups:
- Standard Dose Group: 50 ug dose of mRNA-1273
- Mid Dose Group: 100 ug dose of mRNA-1273
Period: Overall Study
Arm/Group | Standard Dose Group | Mid Dose Group
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was unable to progress beyond the first cohort, and as a result, the high-dose sentinel group did not commence.
Groups:
- Standard-dose - Initial Group: 50 ug ) mRNA-1273 booster vaccine
- Mid-dose - Sentinel Group: 100 ug ) mRNA-1273 booster vaccine
- High-dose - Sentinel Group: 200 ug ) mRNA-1273 booster vaccine
- Total: Total of all reporting groups
Arm/Group | Standard-dose - Initial Group | Mid-dose - Sentinel Group | High-dose - Sentinel Group | Total
Number analyzed (Participants) | 8 | 11 | 0 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 0 | 12
  >=65 years | 2 | 5 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 0 | 6
  Male | 6 | 7 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 5
  Not Hispanic or Latino | 3 | 8 | 0 | 11
  Unknown or Not Reported | 2 | 1 | 0 | 3
Count of Participants [Count of Participants; unit: Participants] | 8 | 11 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Solicited Local and Systemic Reactogenicity Adverse Reactions (AR)
Description: Solicited local and systemic reactogenicity adverse events were documented daily in a dedicated diary, and assigned a grade 1-3 according to the "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" (FDA grading scale). Higher grades are assigned to more severe events.
Time Frame: Day 1 - Day 7 after study drug administration
Measure: Number; unit: participants
Groups:
- Standard-dose: mRNA-1273 (Moderna COVID-19 vaccine) 50 ug
  mRNA-1273 (Moderna COVID-19 vaccine): Study Drug administered via intramuscular injection (IM). Only one dose of study drug administered for the study.
- Mid-Dose: mRNA-1273 (Moderna COVID-19 vaccine) 100 ug
  mRNA-1273 (Moderna COVID-19 vaccine): Study Drug administered via intramuscular injection (IM). Only one dose of study drug administered for the study.
Arm/Group | Standard-dose | Mid-Dose
Number analyzed (Participants) | 8 | 11
participants
  Any Local AR | 5 | 9
  Injection site pain -Grade 1 | 4 | 7
  Injection site pain -Grade 2 | 2 | 4
  Injection Site Swelling-Grade 1 | 0 | 1
  Injection site swelling, Grade 2 | 0 | 1
  Any Systemic AR | 3 | 3
  Fatigue - grade 1 | 1 | 1
  Fatigue - Grade 2 | 2 | 1
  Fatigue - Grade 3 | 1 | 1
  Headache - Grade 1 | 2 | 2
  Headache - Grade 2 | 1 | 1
  Headache - Grade 3 | 1 | 0
  Myalgia - Grade 1 | 1 | 1
  Arthralgia - Grade 1 | 1 | 0
  Chills - Grade 1 | 0 | 1
  Nausea/Vomiting - Grade 1 | 1 | 0
  Nausea/Vomiting - Grade 2 | 1 | 0
  Nausea/Vomiting - Grade 3 | 1 | 0

2. Primary Outcome: Participants Reporting Unsolicited Adverse Events (AEs) Recorded on a Daily Diary
Description: Comprehensive recording of occurrence and severity grade of unsolicited adverse events (AEs) daily. These events were documented in a dedicated diary starting from Day 1 of the study and continued through to Day 30. Data collection encompassed adverse events not specifically solicited, with each event's frequency recorded for analysis.
Time Frame: Day 1 - Day 30 after study drug administration
Measure: Count of Participants; unit: Participants
Groups:
- Standard Dose Group: mRNA-1273 (Moderna COVID-19 vaccine) 50 ug
  mRNA-1273 (Moderna COVID-19 vaccine): Study Drug administered via intramuscular injection (IM). Only one dose of study drug administered for the study.
- Mid Dose Group: mRNA-1273 (Moderna COVID-19 vaccine) 100 ug
  mRNA-1273 (Moderna COVID-19 vaccine): Study Drug administered via intramuscular injection (IM). Only one dose of study drug administered for the study.
Arm/Group | Standard Dose Group | Mid Dose Group
Number analyzed (Participants) | 8 | 11
Participants
  Any unsolicited AE | 1 | 7
  Pain in extremity - left foot, Moderate | 0 | 1
  Pain in extremity - bilateral shoulder pain, Mild | 0 | 1
  Fatigue, Mild | 0 | 1
  Fatigue, Moderate | 0 | 1
  Hyperkalemia, Moderate | 0 | 1
  Creatinine increased, Mild | 0 | 1
  COVID-19 infection - Mild | 1 | 2
  COVID-19 infection - Moderate | 0 | 3
  Joint irritation of left foot and left hand, Mild | 0 | 1
  Dyspnea, Mild | 0 | 1
  Palpitations, Mild | 0 | 1
  LE edema, Mild | 0 | 1
  Mitral regurgitation worsening, Severe | 0 | 1
  Chest heaviness, Mild | 1 | 0
  Shortness of breath worsening, Mild | 1 | 0
  Chest discomfort worsening, Mild | 1 | 0
  Lightheadedness, Mild | 0 | 1
  Mechanical trip and fall, Moderate | 0 | 1
  Left flank pain, Moderate | 0 | 1
  Dry cough, Moderate | 0 | 1

3. Primary Outcome: Participants Reporting Any Serious Adverse Experiences (SAEs) and Adverse Events of Special Interests (AESIs) Related to the Intervention From Day 1 Until Day 180.
Description: This comprehensive data collection is intended to provide insights into the occurrence of significant adverse events and specific adverse events of interest over an extended period
Time Frame: Day 1 - Day 180 after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Group | Mid Dose Group
Number analyzed (Participants) | 8 | 11
Participants | 0 | 0

4. Secondary Outcome: Humoral Immunogenicity Measured by Anti-RBD and Anti-spike (S-2P) IgG Levels at Day 30.
Description: This evaluation provides insights into the vaccine's ability to induce an immune response by quantifying specific antibody levels targeting key viral components, contributing to the understanding of vaccine efficacy and immune response dynamics.
Time Frame: Day 30 after study drug administration
Population: We did not run the assay described. The humoral immunogenicity was measured as neutralizing antibodies since the COVID immunogenicity field had progressed and binding antibodies were not being reported in the literature (only the neutralizing antibodies for the most part).
Arm/Group | Standard Dose Group | Mid Dose Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Humoral Immunogenicity Measured by Neutralizing Antibody Titers From a Pseudovirus Neutralization Assay at Day 30.
Description: Provide a direct measure of the vaccine-induced immune response's ability to neutralize viral infection, offering critical insights into vaccine efficacy and immune response effectiveness
Time Frame: Day 1, Day 30 after study drug administration
Measure: Median (Full Range); unit: Titer
Arm/Group | Standard Dose Group | Mid Dose Group
Number analyzed (Participants) | 8 | 11
Titer
  Neutralizing antibody titre - Day 1 | 4260 [57 to 30788] | 6514 [40 to 14825]
  Neutralizing antibody titre - Day 30 | 5436 [40 to 46022] | 5293 [40 to 9791]

6. Secondary Outcome: Cellular Immunogenicity (CD8+ T Cell Responses After Spike Protein Peptide Pool Stimulation) Measured by Cellular Response Assays Including Flow Cytometry With Intracellular Staining.
Description: Percent of total CD8+ T Cells to quantify vaccine-induced cellular immune response, the activation and functionality of specific immune cell populations to contribute to understanding the vaccine's ability to elicit a robust cellular immune response, which is essential for effective protection against viral infections.
Time Frame: Day 1, Day 30 after study drug administration
Measure: Median (Full Range); unit: percent of total CD8+ T Cells detectable
Arm/Group | Standard Dose Group | Mid Dose Group
Number analyzed (Participants) | 8 | 11
percent of total CD8+ T Cells detectable
  Day 1-IFNγ | 0.01 [0.01 to 0.13] | 0.01 [0.01 to 0.82]
  Day 30-IFNγ | 0.04 [0.01 to 0.16] | 0.01 [0.01 to 0.26]
  Day 1-IL-2 | 0.01 [0.01 to 0.10] | 0.01 [0.01 to 0.10]
  Day 30-IL-2 | 0.01 [0.01 to 0.52] | 0.01 [0.01 to 0.52]
  Day 1-TNFα | 0.01 [0.01 to 0.42] | 0.01 [0.01 to 0.02]
  Day 30-TNFα | 0.01 [0.01 to 0.29] | 0.01 [0.01 to 0.58]
  Day 1- IFNγ, IL-2, or TNFα | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.67]
  Day 30-IFNγ, IL-2, or TNFα | 0.01 [0.01 to 0.48] | 0.01 [0.01 to 0.51]

7. Secondary Outcome: Cellular Immunogenicity (CD4+ T Cell Responses After Spike Protein Peptide Pool Stimulation) Measured by Cellular Response Assays Including Flow Cytometry With Intracellular Staining.
Description: Percent of total CD4+ T Cells to quantify vaccine-induced cellular immune response, the activation and functionality of specific immune cell populations to contribute to understanding the vaccine's ability to elicit a robust cellular immune response, which is essential for effective protection against viral infections.
Time Frame: Day 1, Day 30 after study drug administration
Measure: Median (Full Range); unit: percent of total CD4+ T Cells detectable
Arm/Group | Standard Dose Group | Mid Dose Group
Number analyzed (Participants) | 8 | 11
percent of total CD4+ T Cells detectable
  Day 1-IFNγ | 0.01 [0.01 to 0.59] | 0.01 [0.01 to 0.26]
  Day 30-IFNγ | 0.04 [0.01 to 0.65] | 0.02 [0.01 to 0.20]
  Day 1-IL-2 | 0.01 [0.01 to 0.53] | 0.07 [0.01 to 1.93]
  Day 30-IL-2 | 0.05 [0.01 to 0.31] | 0.20 [0.01 to 0.99]
  Day 1-TNFα | 0.03 [0.01 to 0.62] | 0.01 [0.01 to 0.37]
  Day 30-TNFα | 0.15 [0.01 to 0.95] | 0.01 [0.01 to 0.17]
  Day 1- IFNγ, IL-2, or TNFα | 0.01 [0.01 to 0.43] | 0.01 [0.01 to 0.34]
  Day 30-IFNγ, IL-2, or TNFα | 0.23 [0.01 to 1.13] | 0.01 [0.01 to 0.29]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study, Visit 1 (Day 1) through Visit 6 (Day 180)
Description: The High Dose Group did not have any enrolled participants in this study. This decision was influenced by the availability of the vaccine to the public starting in September 2022. Therefore, results for this arm/group are not reported
Arm/Group | Standard-dose | Mid-Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/11
Other Adverse Events (participants affected / at risk) | 5/8 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard-dose (N=8) | Mid-Dose (N=11)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID 19 infection (Infections and infestations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Post-aspiration pneumonia dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post-op chest paqin (General disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mitral valve regurgitation (MR) and aortic valve regurgitation (AR) post valve replacement surgery (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard-dose (N=8) | Mid-Dose (N=11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest heaviness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
COVID 19 infection (Infections and infestations) | 1 (1) | 4 (5)
Increased Creatinine (General disorders) | 0 (0) | 1 (1)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (4) | 4 (5)
Headache (General disorders) | 3 (5) | 3 (3)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 5 (6) | 10 (12)
Injection site swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Joint irritation, foot and hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Edema of lower extremity (Vascular disorders) | 0 (0) | 1 (1)
Flank pain, left (General disorders) | 0 (0) | 1 (1)
Lightheadedness (General disorders) | 0 (0) | 1 (1)
Mechanical trip and fall (General disorders) | 0 (0) | 1 (1)
Myalgia (General disorders) | 1 (1) | 1 (1)
Nausea/Vomiting (General disorders) | 1 (3) | 0 (0)
Pain in extremity - bilateral shoulder (General disorders) | 0 (0) | 1 (1)
Pain in extremity - left foot (General disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Chest discomfort worsening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of breath worsening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mitral regurgitation worsening (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT05280158/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT05280158/ICF_001.pdf